CLINICAL TRIAL: NCT01082276
Title: Rifampin Drug-Drug Interaction Study With Lurasidone HCl
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D1050270
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Male, Healthy Normal Subjects
Keywords: Rifampin DDI with Lurasidone HCl
MeSH Terms: interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rifampin/Lurasidone (Other): Healthy Normal Subject
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: Lurasidone HCl — 40mg, Single-dose of lurasidone 40 mg (one 40 mg tablet) on Day 1. Daily dosing of rifampin 600 mg (two 300 mg capsules) on Days 1-8. On Day 8, subjects will also receive a single-dose of lurasidone 40 mg (one 40 mg tablet).

SUMMARY:
The effect of rifampin on the pharmacokinetics of lurasidone

DETAILED DESCRIPTION:
by performing an open-label, 2-period, sequential study in healthy subjects. All subjects (N=20) will be assigned to the same treatment sequence, 40 mg po dosing.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects must be of nonchildbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or post-menopausal ≥ 1 year) with follicle stimulating hormone [FSH] > 40 U/L).
2. Subjects with partners of child-bearing potential must agree to use barrier contraception during the study and for 90 days after discharge. Volunteers must agree to not donate sperm during the study and for 90 days after discharge.

Exclusion Criteria:

1. Any disorder that would interfere with the absorption, distribution, metabolism, or excretion of drugs.
2. Use of concomitant medications that prolong the QT/QTc interval from 14 days prior to day - 2 to discharge.
3. Use of any inhibitor or inducer of CYP3A4 taken within 30 days prior to study Day -2
4. Use of (an) investigational drug(s) within the 30 days or 5 half-lives (whichever was longer) prior to Screening.
5. Previous exposure to lurasidone (SM-13496).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — PAREXEL Clinical Pharmacology Research Unit at Baltimore, MD
Locations (1):
- PAREXEL Clinical Pharmacology Research Unit, Baltimore, Maryland, United States